CLINICAL TRIAL: NCT05659680
Title: Achieving Conduction System Activation With Leadless Left Ventricular Endocardial Pacing
Acronym: ACCESS-CRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307507
Record Dates: First submitted 2022-10-18; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac resynchronisation therapy; leadless pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leadless Conduction System Pacing (Experimental): Participants receive leadless conduction system pacing using the WiSE-CRT device.
  Interventions: Device: WiSE-CRT

INTERVENTIONS:
Device: WiSE-CRT — Participants undergo pre-procedural CT, implantation of the WiSE-CRT system targeting the left bundle branch area, and post procedural non-invasive electro-anatomical mapping using electrocardiographic imaging and haemodynamic assessment.
  Other Names: WiSE CRT

SUMMARY:
The goal of this prospective non-randomised study is to test the feasibility of leadless conduction system pacing using the WiSE-CRT device in patients with an indication for Cardiac Resynchronisation Therapy.

The main question[s] it aims to answer are:

1. What is the safety profile of leadless conduction system pacing?
2. What is the success rate of leadless conduction system pacing?
3. What are the electrical and haemodynamic effects of leadless conduction system pacing.

Participants will undergo pre-procedural cardiac CT, and post-procedure electro-anatomical mapping and haemodynamic assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Ability to provide informed consent to participate and willing to comply with the clinical investigation plan and follow-up schedule.
* Patients meeting European Society of Cardiology Criteria for Cardiac Resynchronization Therapy (CRT) with Class 1 or 2a recommendation:

  * Dyssynchronous Heart Failure: Left Ventricular Ejection Fraction (LVEF) ≤35%, QRS duration >150ms or >130ms in presence of left bundle branch block (LBBB). Also included here are patients with EF ≤35%, an existing pacing system and an RV pacing burden of >20%.
  * BLOCK HF population: Patients requiring pacing for atrioventricular (AV) block with an LVEF ≤50%
  * AV node ablation (AVNA) population: Patients planned for AVNA with EF ≤50%.

Exclusion Criteria:

* Any contraindication to LV endocardial pacing.

  * LV thrombus
  * Contra-indication to heparin
  * Contra-indication to anti-platelet agents
* Failure of acoustic window screening
* Septal wall thickness <5mm (minimum required wall thickness at any target implant site)
* Myocardial infarction within 40 days prior to enrolment.
* Cardiac surgery or coronary revascularisation procedure within 3 months prior to enrolment or to be scheduled for such procedures within the following 7 months.
* Participation in other studies with active treatment/investigational arm.
* Pregnant or planning to become pregnant in the next 7 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Procedure/Device related complication rate | 6 months
  Number of procedure or device related complications

SECONDARY OUTCOMES:
Success rate | 6 months
  Percentage of successful tracking
LV function | 6 months
  Percentage of patients with a 15% reduction in LV end systolic volume
Clinical outcome | 6 months
  Percentage of patients with improvement in NYHA class
ECG outcome | 6 months
  Mean change in QRS duration
Biventricular activation time | 6 weeks
  Mean change in biventricular activation time
Haemodynamic improvement | 6 weeks
  Mean change in acute haemodynamic dP/dT

IPD SHARING:
Plan to Share IPD: No